CLINICAL TRIAL: NCT06051188
Title: Flow Versus Pressure Controlled Ventilation in Patients With Moderate to Severe Acute Respiratory Distress Syndrome
Brief Title: FCV vs PCV in Moderate to Severe ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Henrik Endeman, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABR NL83234.078.23
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Distress Syndrome; Ventilator Lung
Keywords: Flow-controlled ventilation; ARDS; Electrical Impedance Tomography; Mechanical Power
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized crossover physiological pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCV-PCV (Experimental): 90 minutes of flow-controlled ventilation followed by 90 minutes of pressure-controlled ventilation.
  Interventions: Device: Flow-controlled ventilation
- PCV-FCV (Experimental): 90 minutes of pressure-controlled ventilation followed by 90 minutes of flow-controlled ventilation.
  Interventions: Device: Flow-controlled ventilation

INTERVENTIONS:
Device: Flow-controlled ventilation — Flow-controlled ventilation (FCV)

SUMMARY:
The goal of this clinical trial is to compare flow-controlled ventilation (FCV) and pressure-controlled ventilation (PCV) in patients with moderate to severe acute respiratory distress syndrome on the intensive care unit.

The main questions it aims to answer are:

* Is the mechanical power during flow-controlled ventilation lower than during pressure-controlled ventilation
* To gain more understanding about other physiological effects and potential benefits of flow-controlled ventilation in comparison to pressure-controlled ventilation (o.a. the end-expiratory lung volume and homogeneity of ventilation).

Participants will be randomized between two ventilation mode sequences, being 90 minutes of FCV followed by 90 minutes of PCV or vice versa.

DETAILED DESCRIPTION:
Rationale: During controlled mechanical ventilation (CMV) only the inspiration is controlled by either a set driving pressure (Pressure Controlled Ventilation, PCV) or tidal volume (Volume Controlled Ventilation, VCV). The expiration depends on the passive elastic recoil of the respiratory system and cannot be controlled and lasts until the airway pressure is equal to the positive end-expiratory pressure (PEEP). The exponential decrease in airway pressure during expiration may result in alveolar collapse and hypoxemia. Flow controlled ventilation (FCV) is a mechanical ventilation method that uses a constant flow during both inspiration and expiration. FCV results in a gradual decrease in airway pressure during expiration as flow is controlled. In both animal and prospective crossover studies, controlled expiration resulted in higher mean airway pressures with reduced alveolar collapse. Besides, FCV resulted in a higher ventilation efficiency measured by a decrease in minute volume at stable arterial partial pressures of carbon dioxide (PaCO2). Where a reduction in alveolar collapse may lead to less atelectrauma, a higher ventilation efficiency may lead to a lower mechanical power (MP), which is the amount of energy (Joules) that is transferred to the respiratory system by the mechanical ventilator every minute. Both are important determinants of Ventilator Induced Lung Injury (VILI). This makes FCV a very interesting ventilation mode in patients with the acute respiratory distress syndrome (ARDS) in which VILI is still a major contributor to overall morbidity and mortality. Two prior prospective cross-over studies have been performed in (COVID-19) ARDS patients that did show a lower minute volume with FCV compared to PCV or VCV. However, these studies did not take into account assessments of the MP or end-expiratory lung volume (EELV), which is a measurement of lung aeration.

The investigators hypothesize that FCV in patients with moderate to severe ARDS results in a lower MP and an increased EELV compared to standard CMV modes (PCV or VCV).

Objectives: To study the effect of FCV on the MP and the EELV compared to PCV.

Study design: Randomized crossover physiological pilot study comparing FCV and PCV.

Study population: Patients with moderate to severe ARDS ≥ 18 years old receiving CMV.

Intervention: Patients are mechanically ventilated with PCV mode at baseline. Upon inclusion the EIT-belt and an esophageal balloon are placed to assess the EELV and transpulmonary pressures respectively. Besides, participants are randomized between the sequence of ventilation mode, namely 90 minutes of PCV followed by 90 minutes of FCV or 90 minutes of FCV followed by 90 minutes of PCV. When PCV is switched to FCV the same mechanical ventilator settings are used as in the PCV mode. After half an hour on FCV the PEEP, driving pressure and flow of FCV are optimized based on the highest compliance and lowest flow matching with a stable PaCO2 thereby not exceeding lung protective ventilation limits (transpulmonary driving pressure ≤ 12cmH2O and tidal volumes ≤ 8 ml/kg ideal body weight (IBW)). PCV is always set according to standard of care. Total time of measurements / study time is 180 minutes.

Main study parameters/endpoints: Primary endpoint is the difference in MP after 90 minutes on FCV compared to after 90 minutes of PCV. An important secondary endpoint is the difference in EELV after 30 minutes on FCV compared to after 30 minutes of PCV.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participants are sedated and on CMV, therefore there will be no discomfort for the patient. FCV has been successfully applied during surgery and on the ICU and the patient will be monitored continuously so the clinical team can act directly in case of any adverse event. Lung volume is measured with EIT, a non-invasive, radiation-free monitoring tool. Transpulmonary pressures are measured with an esophageal balloon that is placed in a similar manor as a nasogastric feeding tube. During optimization of FCV no lung protective ventilation limits will be exceeded. Therefore, overall, the risks of this study are limited.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Provided written informed consent
* Undergoing controlled mechanical ventilation via an endotracheal tube
* Meeting all criteria of the Berlin definition of ARDS

  * Hypoxic respiratory failure within 1 week of a known clinical insult or new or worsening respiratory symptoms
  * Bilateral opacities on X-ray or CT-scan not fully explained by effusions, lobar/lung collapse (atelectasis), or nodules
  * Respiratory failure not fully explained by cardiac failure or fluid overload.
  * Oxygenation: moderate ARDS P/F ratio between 101-200 mmHg, severe ARDS PF ratio ≤ 100mmHg, both with PEEP ≥ 5 cmH2O.
* Intubated ≤72 hours

Exclusion Criteria:

* Severe sputum stasis or production requiring frequent bronchial suctioning (more than 5 times per nurse shift)
* Untreated pneumothorax (i.e., no pleural drainage)
* Hemodynamic instability defined as a mean arterial pressure below 60mmHg not responding to fluids and/or vasopressors or a noradrenalin dose >0.5mcrg/kg/min
* High (>15 mmHg) or instable (an increase in sedation or osmotherapy is required) intracranial pressure
* An inner tube diameter of 6mm or less
* Intubated > 72 hours
* Anticipating withdrawal of life support and/or shift to palliation as the goal of care
* Inability to perform adequate electrical impedance tomography (EIT) measurements with, e.g.:

  * Have a thorax circumference inappropriate for EIT-belt
  * Thoracic wounds, bandages or deformities preventing adequate fit of EIT-belt
  * Recent (<7 days) pulmonary surgery including pneumonectomy, lobectomy or lung transplantation
  * ICD device present (potential interference with proper functioning of the EIT device and ICD device)
  * Excessive subcutaneous emphysema
* Contra-indications for nasogastric tube or inability to perform adequate transpulmonary pressure measurements with, e.g.:

  * Recent esophageal surgery
  * Prior esophagectomy
  * Known presence of esophageal varices
  * Severe bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mechanical power | 90 minutes
  Difference in mechanical power in J/min after 90 minutes of flow-controlled ventilation and 90 minutes of pressure-controlled ventilation

SECONDARY OUTCOMES:
End-expiratory lung volume | 30 minutes
  Difference in end-expiratory lung volume in milliliters after 30 minutes of flow-controlled ventilation and 30 minutes of pressure-controlled ventilation
Dissipated energy | 90 minutes
  Difference in dissipated energy in J/L after 90 minutes of flow-controlled ventilation and 90 minutes of pressure-controlled ventilation
Airway pressures | 30 and 90 minutes
  Difference in airway pressures in cmH2O (PEEP, PEEPtotal, Ppeak, Pplateau, Pdrive) between FCV and PCV
Transpulmonary pressures | 30 and 90 minutes
  Difference in transpulmonary pressures in cmH2O (end-inspiratory transpulmonary pressure, end-expiratory transpulmonary pressure and transpulmonary drivepressure) between FCV and PCV
Minute volume | 30 and 90 minutes
  Difference in minute volume in L/min between FCV and PCV
Ventilatory ratio | 30 and 90 minutes
  Difference in ventilatory ratio between FCV and PCV
Electrical Impedance Tomography (EIT) | 30 and 90 minutes
  Difference in EIT measurements between FCV and PCV (o.a. homogeneity of ventilation)
P/F ratio | 30 and 90 minutes
  Difference in P/F ratio between FCV and PCV
Mean arterial pressure | 30 and 90 minutes
  Difference in mean arterial pressure (mmHg) between FCV and PCV
Pulserate | 30 and 90 minutes
  Difference in pulserate (x/min) between FCV and PCV

CONTACTS AND LOCATIONS:
Overall Officials: Rik Endeman, Dr, Principal Investigator — Erasmus Medical Center
Locations (1):
- Maasstad Hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Oosten JP, Francovich JE, Weller D, Rietdijk W, Goedendorp N, Somhorst P, den Uil CA, Gommers D, Jonkman AH, Endeman H. Flow-controlled ventilation versus pressure-controlled ventilation in moderate to severe ARDS patients: a randomized crossover physiological study. Intensive Care Med Exp. 2025 Dec 24;13(1):137. doi: 10.1186/s40635-025-00847-4. PMID 41442110